CLINICAL TRIAL: NCT05047679
Title: The Effectiveness of Pain Neuroscience Education in Patients at Risk for Unfavorable Outcome Following Surgery for Lumbar Radiculopathy: A Multicentric Randomized Controlled Trial
Brief Title: The Effectiveness of Pain Neuroscience Education in At-risk Patients Following Surgery for Lumbar Radiculopathy
Acronym: B²EARS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues that could not be resolved in a timely manner.
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Jo Nijs, Professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FWOSB108; 1S61521N (Other Grant/Funding Number: Fonds Wetenschappelijk Onderzoek - Vlaanderen (FWO))
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Lumbar Radiculopathy
Keywords: Biomedical Education; Pain Neuroscience Education; Lumbar surgery; Education; Chronic pain; Kinesiophobia; Catastrophization; Perioperative Education
MeSH Terms: conditions — Radiculopathy; Chronic Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the participant and the person responsible for the monitoring of the baseline and follow-up assessments will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative Pain Neuroscience Education (Experimental): Patients in the experimental treatment group will receive Perioperative Pain Neuroscience Education, including a preoperative session 3 days before the surgery, access to an educational web application and a postoperative session 2 days following the surgery. Both education sessions will be face-to-face and will last approximately 60 minutes.
  Interventions: Behavioral: Perioperative Pain Neuroscience Education
- Perioperative Biomedical Education (Active Comparator): Patients in the control treatment group will receive Perioperative Biomedical Education, including a preoperative session 3 days before the surgery, access to an educational web application and a postoperative session 2 days following the surgery. Both education sessions will be face-to-face and will last approximately 60 minutes.
  Interventions: Behavioral: Perioperative Biomedical Education

INTERVENTIONS:
Behavioral: Perioperative Pain Neuroscience Education — Perioperative pain neuroscience education addresses modifiable preoperative risk factors, and in particular cognitive and emotional risk factors, such as fear of movement and pain catastrophizing (i.e., excessively negative orientation toward pain). This education is a cognitive-based therapeutic intervention which reconceptualizes pain, informs patients about what to expect from the evolution of their pain, de-emphasizes the patho-anatomical content and focuses on factors contributing to the development of pain. It explains this all within a biopsychosocial framework, which means that it aims to optimize patients' beliefs. Furthermore, it intends to reassure the patient about the decision to have surgery, to potentially decrease perioperative distress.
  Other Names: Pain Education
  Arms: Perioperative Pain Neuroscience Education
Behavioral: Perioperative Biomedical Education — Perioperative biomedical education will discuss the anatomy, physiology and biomechanics of the lumbar spine with the patient. Additionally, the content of this education includes the expected course of postoperative back and leg pain, as well as ergonomic advice on patient-specific daily activities. This education will be given within a biomedical framework, which means that it aims to explain the patients' complaints and recovery while focusing on anatomy and biomechanics, as opposed to patients' beliefs and cognitions.
  Arms: Perioperative Biomedical Education

SUMMARY:
This study aims to assess the effectiveness of perioperative pain neuroscience education (PPNE) in patients who are at risk for unfavorable outcome following surgery for lumbar radiculopathy. Although most of these surgeries are successful, 23-28% of patients report chronic pain and disability following surgery. Many preoperative factors are associated with an unfavorable surgical outcome, including maladaptive cognitive and emotional factors. Yet, current preoperative education, which focuses on anatomy and biomechanics of the lumbar spine, is ineffective in changing those maladaptive factors. PPNE was introduced as an innovative therapy that addresses modifiable risk factors in patients undergoing surgery for lumbar radiculopathy. PPNE reconceptualizes pain, informs patients about their pain development and is well established for improving maladaptive cognitions in several chronic pain-populations. Hence, we hypothesize that PPNE will be more effective than perioperative biomedical education in improving postsurgical quality of life, pain, analgesic use and return to work in patients at risk for unfavorable outcome following surgery for lumbar radiculopathy. First, a multicentric randomized controlled trial will compare the therapy effects of PPNE to perioperative biomedical education in these at-risk patients. Next, the mediating role of changes in maladaptive cognitions, such as fear of movement and pain catastrophizing, on the therapy effect of PPNE will be investigated.

DETAILED DESCRIPTION:
Study rationale: Lumbar radiculopathy is described as uni- or bilateral leg pain which is often worse than back pain, with pain radiating in the related dermatomes and possible associations with sensory and/or motor symptoms or even deficits. Although surgical intervention for lumbar radiculopathy is often considered anatomically successful, several patients undergoing similar surgeries continue to experience pain and disability. Furthermore, patients developing such an unfavorable outcome also report decreased quality of life values, as well as an increase in analgesic use and health care utilization. Such unfavorable outcome is associated with a multitude of preoperative factors, including but not limited to maladaptive cognitive and emotional factors (e.g., fear of movement, pain catastrophizing, anxiety, distress and depression), preexisting chronic pain and long duration of preoperative sick leave. In line with this, it has been suggested that maladaptive psychological factors require special attention and optimization before surgery. Perioperative pain neuroscience education (PPNE) is such an intervention addressing these maladaptive psychological factors, such as fear of movement and pain catastrophizing. Therefore, a study assessing the effectiveness of PPNE on surgical outcome in at-risk patients undergoing surgery for lumbar radiculopathy is warranted.

Rationale for study design: The present study builds on the evidence provided by the study of Louw et al. (2014 & 2016) which was a randomized controlled trial comparing PPNE with no supplemental intervention in patients undergoing surgery for lumbar radiculopathy. As such, we will conduct a multicentric randomized controlled trial investigating the therapy effect of PPNE specifically in patients with lumbar radiculopathy at risk for unfavorable surgical outcome. Doing this we will address several knowledge gaps by comparing two balanced therapy groups (PPNE vs perioperative biomedical education (PBE)), therefore overcoming potential bias due to unbalanced treatment arms, by adding several relevant outcome measures, and by targeting high-risk patients rather than all patients undergoing surgery.

Study objectives: The primary objective is to examine whether PPNE is more effective than PBE in improving postoperative quality of life at 6 weeks follow-up in patients undergoing surgery for lumbar radiculopathy at risk for unfavorable surgical outcome. Secondary objectives include: 1) to explore baseline associations between pain cognitions, quality of life and pain in patients scheduled for surgery for lumbar radiculopathy at risk for unfavorable outcome; 2) to examine whether PPNE is more effective than PBE in obtaining good surgical results concerning quality of life, pain, analgesic use, return to work, self-reported symptoms of central sensitization and pain cognitions at 6 weeks, 6 months and 1 year post-surgery and 3) to reveal the mediating role of changes in pain cognitions in the mechanism behind the therapy effect of PPNE in patients undergoing surgery for lumbar radiculopathy at risk for unfavorable outcome.

Study design: This study is a randomized controlled trial with one-year follow-up using preoperative patient screening based on chronic pain (≥ 6 months), kinesiophobia (Tamp Scale for Kinesiophobia ≥ 37/68) and pain catastrophizing (Pain Catastrophizing Scale ≥ 30/52). Eligible patients undergoing surgery for lumbar radiculopathy will be randomized and receive either the experimental intervention, i.e., PPNE, or the control intervention, i.e., PBE. Follow-up assessments will be organized at 6 weeks, 6 months and 12 months following the surgery.

Patient recruitment: All patients scheduled for surgery for lumbar radiculopathy in one of the participating hospitals will be contacted by telephone by the coordinating investigator. First, patients will be informed about the project and asked if they are willing to participate. When patients agree with participating in the study, they will be screened for potential eligibility using the in- and exclusion criteria. Following the initial screening, patients will have to meet an additional set of presurgical criteria (i.e., chronic pain, pain catastrophizing and kinesiophobia) to assess whether they are at risk for unfavorable surgical outcome, and therefore eligible for inclusion in the study sample. To screen for these presurgical criteria, patients eligible for further screening after the initial telephone interview, will be asked to complete an online survey questioning the three aforementioned criteria. The first page of the online survey will inform the patients once again about the goal of the screening and all patients will have to indicate their consent (by checking a box) before they can proceed to the actual questionnaire.

Randomization and blinding procedures: Following baseline assessments, participants will be randomized to one of both treatment groups. Concealed randomization will be prepared using a stratified permuted block allocation with stratification for treatment center. Randomization will be executed by an independent researcher who is not involved in the recruitment, assessments, treatment provision or statistical analyses. Patients will not know whether the intervention they receive is the experimental or the control intervention, however they will of course be aware of the content of the received intervention. A co-investigator, who will be responsible for baseline assessment and all follow-up assessments, will also be blinded to group allocation. With regard to this, patients will be asked not to communicate with the co-investigator about the intervention they received. The therapists providing the experimental treatment will not be involved in providing the control intervention and vice versa.

Sample size: Sample size was calculated to be 108 (54 per intervention group) based on a medium effect size of 0.6, α of 0.05, desired power of 0.80, an allocation ratio (N2/N1) of 1 and an anticipated loss to follow-up of 20%. A longitudinal pilot study in patients undergoing surgery for lumbar radiculopathy and who were retrospectively selected based on chronic pain (≥3 months), kinesiophobia (Tampa Scale for Kinesiophobia ≥37/68) and pain catastrophizing (Pain Catastrophizing Scale ≥30/52) was performed and evaluated the effect of PPNE on Short-Form 36-item, these results were used to determine the effect size for the sample size calculation.

Statistical analysis: Descriptive and correlation analyses will be performed on the baseline data. An AN(C)OVA repeated measures analysis will be used to evaluate treatment effects (primary and secondary objective). Lastly, a mediation analysis will be performed to examine the potential mediating role of changes in pain cognitions on the therapy effect of PPNE on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgery for lumbar radiculopathy
* Aged 18 years or older
* Willing to comply with pre-determined follow-up
* Speaking and reading Dutch fluently
* No new treatments/medication 3 weeks prior to participation and during the trial
* Having chronic back and/or leg pain ≥ 6 months
* Scoring ≥ 37/68 on the Tampa Scale for Kinesiophobia
* Scoring ≥ 30/52 on the Pain Catastrophizing Scale

Exclusion Criteria:

* Surgery for another condition
* Symptoms of cord compression or bilateral leg pain
* Other chronic illness characterized by chronic pain
* Other chronic rheumatoid, neurological, endocrinological, psychiatric or cognitive disorders
* Indicated cognitive impairment (Scoring ≤11/15 on the 5-min Telephone Montreal Cognitive Assessment)
* Pregnant or have given birth during the past year
* No access to computer, or mobile device at home
* Complications during the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life | Change between baseline (1 week before surgery) and 6 weeks post-surgery, baseline and 6 months post-surgery, baseline and 1 year post-surgery*
  Change in health-related quality of life will be be assessed by the Short Form 36-item Health Survey (SF-36). The SF-36 contains 8 subscales: physical, emotional, social and role functioning, bodily pain, mental health, vitality and general health. The psychometric properties are well established in a wide variety of patient populations, and its responsiveness to change following surgical interventions is superior than other generic health status measurement scales commonly used in evaluations of interventions for chronic, disabling pain. Additionally, the 5-level EuroQol 5-dimensions (EQ-5D*), which also has good measurement properties, will be used to calculate the change in health utility values between baseline and 1 year post-surgery.

SECONDARY OUTCOMES:
Change in self-reported leg and low back pain intensity | Change between baseline (1 week before surgery) and 6 weeks post-surgery, baseline and 6 months post-surgery, baseline and 1 year post-surgery
  Pain intensity for the leg and low back will be assessed by a series of 100mm Visual Analogue Scales (VAS). The VAS pain score is believed to be reliable, valid and sensitive to change. More specifically the patient will be asked to rate their highest and lowest pain severity in the last 24 hours for back or leg pain, and mean pain in the last 24 hours, as well as current pain for the back and leg separately.
Change in analgesic use | Change between baseline (1 week before surgery) and 6 weeks post-surgery, baseline and 6 months post-surgery, baseline and 1 year post-surgery
  Analgesic use will be assessed by a self-reported recall questionnaire, which has been proven to be valid and feasible for a period up to 6 months. Patients will be asked to report the name of the medication, frequency of use, dose and whether it was prescribed or not. Also, patients are asked to indicate whether the medication was taken because of their back or leg pain, and if not, what the reason was for taking this medication.
Return to work (6 weeks post-surgery) | 6 weeks post-surgery
  Return to work will be assessed by asking patients whether they already resumed professional activities, and if yes, since when they resumed work and to what extent. Also, patients will be given the opportunity to mention whether they had to change jobs or job content for effective work resumption. Additionally, prescribed sick leave is recorded separately by asking patients to report the dates of the doctor's notes.
Return to work (6 months post-surgery) | 6 months post-surgery
  Return to work will be assessed by asking patients whether they resumed or maintained professional activities, and if yes, since when they resumed work and to what extent they are currently working. Also, patients will be given the opportunity to mention whether they had to change jobs or job content for effective work resumption or maintenance. Additionally, prescribed sick leave is recorded separately by asking patients to report the dates of the doctor's notes.
Return to work (1 year post-surgery) | 1 year post-surgery
  Return to work will be assessed by asking patients whether they resumed or maintained professional activities, and if yes, since when they resumed work and to what extent they are currently working. Also, patients will be given the opportunity to mention whether they had to change jobs or job content for effective work resumption or maintenance. Additionally, prescribed sick leave is recorded separately by asking patients to report the dates of the doctor's notes.
Change in self-reported symptoms of central sensitization | Change between baseline (1 week before surgery) and 6 weeks post-surgery, baseline and 6 months post-surgery, baseline and 1 year post-surgery
  The Dutch Central Sensitization Inventory (CSI) will be used to assess self-reported symptoms of central sensitization. The CSI consists of 25 statements about symptoms that people with chronic pain might encounter, such as sensitivity to light or concentration difficulties. A reported higher degree of self-symptomology regarding central sensitization indicates the potential presence of hypersensitivity. It shows good validity for assessing symptoms of central sensitization in patients with chronic pain.
Change in kinesiophobia | Change between baseline (1 week before surgery) and 6 weeks post-surgery, baseline and 6 months post-surgery, baseline and 1 year post-surgery
  Kinesiophobia will be assessed with the Tampa Scale for Kinesiophobia (TSK), which is a questionnaire consisting of 17 items, and the total score can range from 17 to 68 with higher scores indicating higher levels of kinesiophobia. It has good clinimetric properties in patients with low back pain.
Change in pain catastrophizing | Change between baseline (1 week before surgery) and 6 weeks post-surgery, baseline and 6 months post-surgery, baseline and 1 year post-surgery
  Pain catastrophizing will be assessed with the Pain Catastrophizing Scale (PCS), which has well-established clinimetric properties. It consists of 13 items describing different thought and feelings that individuals may experience when they are experiencing pain, total scores range from 0 to 52, with higher scores indicating more catastrophizing.
Change in pain hypervigilance | Change between baseline (1 week before surgery) and 6 weeks post-surgery, baseline and 6 months post-surgery, baseline and 1 year post-surgery
  Pain hypervigilance will be assessed using the Pain Vigilance and Awareness Questionnaire (PVAQ), which is designed to measure attention to pain by assessing awareness, consciousness, vigilance and observation of pain. This questionnaire consists of 16 items and total scores can range from 0 to 90, with higher scores indicating more pain vigilance. These items have demonstrated good internal consistency reliability (Cronbach's alpha = 0.86) in patients with chronic low back pain.

OTHER OUTCOMES:
Demographic data | Baseline (1 week before surgery)
  Patients will be asked to fulfil a demographic questionnaire concerning their age, gender, height, weight, education level, household composition and professional situation.
Health literacy | Baseline (1 week before surgery)
  Health literacy will be evaluated using the 16-item questionnaire from the Health Literacy Study Europe (HLS-EU-Q16). The HLS-EU-Q16 is the short form of the HLS-EU-Q47, as developed during the European Health Literacy Survey (HLS-EU). The total score is calculated as the sum of all dichotomized answers ('fairly' or 'very' easy = 1; 'fairly' or 'very' difficult = 0) and ranges between 0 and 16. Correlations between the results of the HLS-EU-Q16 and the HLS-EU-Q47 were found to be high and the clinimetric properties of the short form are considered to be acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel
Locations (4):
- Belgium (4):
  - AZ Rivierenland, Bornem, Antwerpen
  - AZ Sint-Dimpna, Geel, Antwerpen
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - ZNA Middelheim, Antwerp

IPD SHARING:
Plan to Share IPD: Yes
Given the confidential nature of the collected data, the raw data will not be made open access following the study. However, excluding all possible personal identifiable data (e.g., date of birth and date of surgery), the pseudonymized data of all outcome measures (i.e., health-related quality of life, pain intensity, analgesic use, return to work, self-reported symptoms of central sensitization, pain catastrophizing, kinesiophobia and pain hypervigilance), as well as general demographic data (e.g., age, height, weight and education level) will be made available via a data repository with restricted access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following the study, the data will be stored at a data repository with restricted access for 10 years.
Access Criteria: Only researchers who intend to use and analyze the pseudonymized data for the purpose of scientific research can request access to the data. Additionally, researchers who intend to use the data are required to provide a statistical plan including the predetermined research question and detailing the intended analyses. Also, details regarding the storage of the shared data should be provided to ensure that the researchers took the appropriate measures to establish a secure storage location for the shared data. A request for data access can be send to the central contact person and a data sharing agreement will be signed by both parties.

REFERENCES:
- [Background] Ickmans K, Moens M, Putman K, Buyl R, Goudman L, Huysmans E, Diener I, Logghe T, Louw A, Nijs J. Back school or brain school for patients undergoing surgery for lumbar radiculopathy? Protocol for a randomised, controlled trial. J Physiother. 2016 Jul;62(3):165. doi: 10.1016/j.jphys.2016.05.009. Epub 2016 Jun 11. PMID 27298051
- [Background] Louw A, Butler DS, Diener I, Puentedura EJ. Development of a preoperative neuroscience educational program for patients with lumbar radiculopathy. Am J Phys Med Rehabil. 2013 May;92(5):446-52. doi: 10.1097/PHM.0b013e3182876aa4. PMID 23478459
- [Background] Louw A, Diener I, Landers MR, Puentedura EJ. Preoperative pain neuroscience education for lumbar radiculopathy: a multicenter randomized controlled trial with 1-year follow-up. Spine (Phila Pa 1976). 2014 Aug 15;39(18):1449-57. doi: 10.1097/BRS.0000000000000444. PMID 24875964
- [Background] Wilson CA, Roffey DM, Chow D, Alkherayf F, Wai EK. A systematic review of preoperative predictors for postoperative clinical outcomes following lumbar discectomy. Spine J. 2016 Nov;16(11):1413-1422. doi: 10.1016/j.spinee.2016.08.003. Epub 2016 Aug 4. PMID 27497886
- [Background] den Boer JJ, Oostendorp RA, Beems T, Munneke M, Oerlemans M, Evers AW. A systematic review of bio-psychosocial risk factors for an unfavourable outcome after lumbar disc surgery. Eur Spine J. 2006 May;15(5):527-36. doi: 10.1007/s00586-005-0910-x. Epub 2005 May 25. PMID 15915334
- [Background] den Boer JJ, Oostendorp RA, Beems T, Munneke M, Evers AW. Continued disability and pain after lumbar disc surgery: the role of cognitive-behavioral factors. Pain. 2006 Jul;123(1-2):45-52. doi: 10.1016/j.pain.2006.02.008. Epub 2006 Mar 24. PMID 16563624
- [Background] Taylor RS, Taylor RJ. The economic impact of failed back surgery syndrome. Br J Pain. 2012 Nov;6(4):174-81. doi: 10.1177/2049463712470887. PMID 26516490
- [Background] Inoue S, Kamiya M, Nishihara M, Arai YP, Ikemoto T, Ushida T. Prevalence, characteristics, and burden of failed back surgery syndrome: the influence of various residual symptoms on patient satisfaction and quality of life as assessed by a nationwide Internet survey in Japan. J Pain Res. 2017 Apr 6;10:811-823. doi: 10.2147/JPR.S129295. eCollection 2017. PMID 28435318
- [Background] Manca A, Eldabe S, Buchser E, Kumar K, Taylor RS. Relationship between health-related quality of life, pain, and functional disability in neuropathic pain patients with failed back surgery syndrome. Value Health. 2010 Jan-Feb;13(1):95-102. doi: 10.1111/j.1524-4733.2009.00588.x. Epub 2009 Aug 20. PMID 19695004
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Truijen S, Craps J, Van den Keybus N, Paul L. Pain neurophysiology education improves cognitions, pain thresholds, and movement performance in people with chronic whiplash: a pilot study. J Rehabil Res Dev. 2011;48(1):43-58. doi: 10.1682/jrrd.2009.12.0206. PMID 21328162
- [Background] Meeus M, Nijs J, Van Oosterwijck J, Van Alsenoy V, Truijen S. Pain physiology education improves pain beliefs in patients with chronic fatigue syndrome compared with pacing and self-management education: a double-blind randomized controlled trial. Arch Phys Med Rehabil. 2010 Aug;91(8):1153-9. doi: 10.1016/j.apmr.2010.04.020. PMID 20684894
- [Background] Louw A, Diener I, Landers MR, Zimney K, Puentedura EJ. Three-year follow-up of a randomized controlled trial comparing preoperative neuroscience education for patients undergoing surgery for lumbar radiculopathy. J Spine Surg. 2016 Dec;2(4):289-298. doi: 10.21037/jss.2016.12.04. PMID 28097246
- [Background] Butler D, Moseley GL. Explain pain: Adelaide: NOI Group Publishing; 2003
- [Background] van Wilgen CP, Nijs J. Pijneducatie: een praktische handleiding voor (para)medici: Bohn Stafleu van Loghum; 2010.
- [Background] Louw A. Your Nerves Are Having Back Surgery. International Spine and Pain Institute, Minneapolis, U.S.A.; 2012.